CLINICAL TRIAL: NCT06116162
Title: Department of Dermatology of Xijing Hospital of Air Force Medicial University
Brief Title: Comparison of SVF-gel Filling and CO2 Fractional Laser on Atrophic Acne Scar Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KY20202029-F-2
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Autologous Fat Graft Harvesting, SVF-gel Preparation and Filling; CO2 Fractional Laser Treatment by Using Acupulse Device

STUDY DESIGN:
Intervention Model Description: Seventeen patients with moderate to severe acne scars were treated with SVF-gel filling and CO2 fractional laser through a 24-week, randomized split-face study. One randomly assigned half side of each patient's received one SVF-gel filling treatment and the other side by two CO2 fractional laser treatment once one months.
Who Masked: Outcomes Assessor
Masking Description: Two dermatologists evaluating the severity of acne scars were blinded to the assignment. At patients' each evaluation visit, photographic assessments by dermatologists, VISIA and Antera 3D analysis and patients' subjective assessments were conducted.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 fractional laser treatment (Active Comparator): One side face was random to receive CO2 fractional laser. After local anesthesia, Acupulse device (LUMENIS, US) was used to perform CO2 fractional laser. The laser was operated in DeepFX mode under the parameters of 20-25 MJ energy intensity, 5% coverage, 300 Hz emission frequency and on the 10 mm spot size without overlap, Superficial mode under the parameters of 80-120 MJ energy intensity, 40-60% coverage, 300 Hz emission frequency, 10 mm spot size without overlap.
  Interventions: Device: SVF-gel Filling and CO2 fractional laser
- SVF-gel preparation and filling (Experimental): The other side face received SVF-gel filling. The autologous fat graft was harvested from the lower abdomen or inner thigh of all subjects. The Coleman fat was was islolated by centrifugation. Then, SVF gel further islolated by using cutting and centrifugation. 22G sharp-tip injector was used to inject the SVF-gel into the dermis of acne scars.
  Interventions: Device: SVF-gel Filling and CO2 fractional laser

INTERVENTIONS:
Device: SVF-gel Filling and CO2 fractional laser — SVF-gel preparation and filling:The autologous fat graft was harvested from the lower abdomen or inner thigh of all subjects. Then the lipoaspirate was centrifuged at 1200g for 3 minutes to obtain Coleman fat in the middle layer. The Coleman fat was then transferred between two syringes until the Coleman fat converted into a uniform emulsion, and then processed by centrifugation at 2000g for 3 min. Finally, the remaining substance under the oil layer was SVF gel. We used a 22G sharp-tip injector to inject the SVF-gel into the dermis of acne scars, and the injected materials were diffusely distributed.
  CO2 fractional laser treatment: After local anesthesia, Acupulse device (LUMENIS, US) was used to perform CO2 fractional laser. The laser was operated in DeepFX mode under the parameters of 20-25 MJ energy intensity, 5% coverage. Superficial mode under the parameters of 80-120 MJ energy intensity, 40-60% coverage.

SUMMARY:
Background Adipose extracellular matrix/stromal vascular fraction gel（SVF-gel）, which contains adipose-derived stem cells, endothelial cells, smooth muscle cells, pericytes, and other cell components.

Objective To determine the efficacy and safety of SVF-gel for treating acne scars and to compare the results with CO2 fractional laser.

Methods Seventeen patients with moderate to severe acne scars were treated with SVF-gel filling and CO2 fractional laser through a 24-week, randomized split-face study. One randomly assigned half side of each patient's received one SVF-gel filling treatment and the other side by two CO2 fractional laser treatment once one months. Clinical improvement was assessed by two blinded investigators with Echelle d'Evaluation Clinique des Cicatrices d'acne (ECCA) scale, VISIA and Antaro-3D detection.

DETAILED DESCRIPTION:
This study was designed as a 24-week, prospective, randomized split-face protocol that compared clinical courses between two facial sides either receiving SVF-gel injection or CO2 fractional laser for acne scars. At the initial presentation, the evaluation of the severity of acne scar by Echelle d'Evaluation Clinique des Cicatrices d'acne (ECCA) scale (Table1), VISIA and Antera 3D analysis for all enrolled patients. Then, each facial side of every patient was randomly assigned into either SVF-gel injection or CO2 fractional laser treatment side. A random allocation sequence was created using computer-based random number generators to assign the treatment modality of each side. Randomization codes were secured in a safe until all data analyses were finished. Each patient was received SVF-gel injection for just one time on one half face, CO2 fractional laser treatment for two consecutive sessions at 8-week intervals on the other half face, with a follow-up visit at 16 weeks after the final CO2 fractional laser treatment. Evaluations of each treatment sessions were performed after 1 week, 2 months of every treatment. Two dermatologists evaluating the severities of acne scars were blinded to the assignment. At patients' each evaluation visit, photographic assessments by dermatologists, VISIA and Antera 3D analysis and patients' subjective assessments were conducted.

ELIGIBILITY:
Inclusion Criteria:

* Acne scar patients with severity of moderate to severe by ECCA scale evaluation.
* All the subjects were not allowed to use any systemic, topical, or light-based acne scar treatment during the course of this study.

Exclusion Criteria:

* pregnancy, mental illness.
* Intake of oral isotretinoin within 3 months
* Application of the other chemical peeling and light-based treatments within 8 weeks

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
ECCA scale score | 3 Month after the second CO2 Fractional Laser treatment
  ECCA scale score of each face before and after the treatment of SVF-gel filling and CO2 Fractional Laser

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Ph.D., Study Director — Xijing Hospital of Air Force University
Locations (1):
- Acupulse device, Xi'an, China

IPD SHARING:
Plan to Share IPD: No
No plan to describe

REFERENCES:
- [Background] Bhargava S, Cunha PR, Lee J, Kroumpouzos G. Acne Scarring Management: Systematic Review and Evaluation of the Evidence. Am J Clin Dermatol. 2018 Aug;19(4):459-477. doi: 10.1007/s40257-018-0358-5. PMID 29744784
- [Background] Connolly D, Vu HL, Mariwalla K, Saedi N. Acne Scarring-Pathogenesis, Evaluation, and Treatment Options. J Clin Aesthet Dermatol. 2017 Sep;10(9):12-23. Epub 2017 Sep 1. PMID 29344322
- [Result] Boen M, Jacob C. A Review and Update of Treatment Options Using the Acne Scar Classification System. Dermatol Surg. 2019 Mar;45(3):411-422. doi: 10.1097/DSS.0000000000001765. PMID 30856634
- [Result] Yao Y, Cai J, Zhang P, Liao Y, Yuan Y, Dong Z, Lu F. Adipose Stromal Vascular Fraction Gel Grafting: A New Method for Tissue Volumization and Rejuvenation. Dermatol Surg. 2018 Oct;44(10):1278-1286. doi: 10.1097/DSS.0000000000001556. PMID 29781904
- [Derived] Zhao T, Li M, Wang J, Liu J, Wei J, Liu X, Gao C, Li B. Comparison of the Effects of Adipose Extracellular Matrix/Stromal Vascular Fraction Gel Injection and CO2 Fractional Laser on Atrophic Acne Scar in Asians Through a 24-Week Prospective, Randomized, Split-Face Study. J Cosmet Dermatol. 2025 Mar;24(3):e70131. doi: 10.1111/jocd.70131. PMID 40112029